CLINICAL TRIAL: NCT05937490
Title: Assisted Reproductive Technology (ART) and Pregnancy Outcomes in Women With Adenomyosis (Internal Endometriosis) According to Stimulation Protocol in Relation to Immunological and Endometrial Features: a Prospective, Randomized Study
Brief Title: Adenomyosis and ART
Acronym: ADENOFERT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Fabio Facchinetti, Head of Obstetrics and Gynecology at the University Hospital unimore, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-2021-12371935
Record Dates: First submitted 2023-06-13; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Adenomyosis
Keywords: Adenomyosis; Assisted reproductive technology; ART
MeSH Terms: conditions — Adenomyosis | interventions — Leuprolide; dienogest; Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Long) (Experimental): COH will be performed using a long GnRH agonist protocol(administration of depot leuprorelin 3.75 mg on day 21 of the previous luteal phase of the stimulation cycle). COH will be commenced when pituitary desensitization was achieved(~14 days after the initiation of GnRH agonists) as evidenced by the absence of ovarian follicles >10 mm and endometrial thickness <4 mm on TV-US examination.
  Interventions: Drug: Enantone
- Group 2 (Long + high dose DNG) (Experimental): Before COH, patients will be treated with DNG at high dose (2 mg+2 mg/day) for 28 days, from the first day of previous menstrual cycle. COH will be performed using a long GnRH agonist protocol (administration of depot leuprorelin 3.75 mg on day 21 of the previous luteal phase of the stimulation cycle). COH will be commenced when pituitary desensitization was achieved (~14 days after the initiation of GnRH agonists), as defined above.
  Interventions: Drug: Dienogest 2 MG (milligram); Drug: Enantone
- Group 3 (ultra-long): (Experimental): COH will be performed using a ultra-long GnRH agonist protocol (administration of the first depot leuprorelin 3.75 mg on day 21 of menstrual cycle, repeated after 28 days for other two times). COH will be commenced when pituitary desensitization was achieved (~14 days after the initiation of GnRH agonists), as described above.
  Interventions: Drug: Enantone
- Control group (without adenomyosis) (Other): COH will be performed by using a long GnRH agonist protocol as previous described or using a flexible GnRH antagonist protocol. During TV-US monitoring, when at least one follicle reached 14 mm in diameter, to achieve LH (luteinizing hormone) suppression avoiding spontaneous ovulation, GnRH antagonist 0.25 mg/day will be added subcutaneously until the day of HCG administration.
  Interventions: Drug: long GnRH agonist or flexible GnRH antagonist protocol.

INTERVENTIONS:
Drug: Enantone — administration of depot leuprorelin 3.75 mg on day 21 of the previous luteal phase of the stimulation cycle.
  Arms: Group 1 (Long)
Drug: Dienogest 2 MG (milligram) — Before COH, patients will be treated with DNG at high dose (2 mg+2 mg/day) for 28 days, from the first day of previous menstrual cycle. COH will be performed using a long GnRH agonist protocol (administration of depot leuprorelin 3.75 mg on day 21 of the previous luteal phase of the stimulation cycle).
  Other Names: Enantone
  Arms: Group 2 (Long + high dose DNG)
Drug: Enantone — COH will be performed using a ultra-long GnRH agonist protocol (administration of the first depot leuprorelin 3.75 mg on day 21 of menstrual cycle, repeated after 28 days for other two times).
  Arms: Group 2 (Long + high dose DNG); Group 3 (ultra-long):
Drug: long GnRH agonist or flexible GnRH antagonist protocol. — During TV-US monitoring, when at least one follicle reached 14 mm in diameter, to achieve LH suppression avoiding spontaneous ovulation, GnRH antagonist 0.25 mg/day will be added subcutaneously until the day of HCG administration.
  Arms: Control group (without adenomyosis)

SUMMARY:
The goal of this clinical trial is to:

* Prospectively investigate the association of Adenomyosis with fertility outcomes in relation to COH protocols for ART (long or ultra- long protocol) with a preventive high-dose anti-inflammatory progestin such as DNG and to assess their association with pregnancy and neonatal outcomes (preterm delivery,pre-eclampsia,Caesarean section,fetal malpresentation,small for gestational age,low birth weight and postpartum hemorrhage).
* Understand how the endometrial interface by studying the response of progesterone and DNG stimulated decidualization markers, correlating them with the success of ART protocol stimulation and to pregnancy specific outcomes
* Evaluate the immune changes during the implantation period and in the different trimesters of the pregnancies after ART conception.

DETAILED DESCRIPTION:
Adenomyosis (internal endometriosis) may negatively influence fertility and perinatal outcomes. Inflammation, immune modulation, oxidative stress, extracellular matrix remodelling, aberrant angiogenesis have been implicated in altered oocyte development, uterine receptivity, implantation, successful maintenance of pregnancy. An improvement for infertile women could be a longer GnRH(gonadotropin-releasing hormone) agonist protocol with the addition of a preventive high-dose progestin treatment during controlled ovarian hyperstimulation (COH) Infertile women with transvaginal ultrasound (TV-US) based diagnosis of adenomyosis treated will be randomized into 3 different protocols of COH. Study group 1: Long COH, Study group 2: Long COH + high-dose dienogest (DNG), Study Group 3: Ultra-long COH. COH in controls without adenomyosis will be performed using a long GnRH agonist protocol as previous described or using a flexible GnRH antagonist protocol, according to clinical practice. Our aim is to include a total of n=250 women with adenomyosis and n=250 healthy women of a similar age and basal features at the first ART attempt. The primary outcome will be the number of live birth defined as delivery of one or more live-born infant at > 22 weeks of gestation. Many secondary outcomes will be evaluated as well.

Subsequent eventual ongoing pregnancies will be followed as in normal clinical practice, in particular for the risk of preterm delivery, pre-eclampsia, Caesarean section, fetal malpresentation,small for gestational age, low birth weight and postpartum hemorrhage. In a subgroup of randomized women, the role of endometrial decidualization and its mechanisms will be evaluated in endometrial cells in vitro looking at the response to progesterone and DNG stimulated decidualization markers (in particular osteopontin and prolactin). The different responses will be related to the outcome of ARt and pregnancy related outcomes (preterm delivery, pre-eclampsia, Caesarean section, fetal malpresentation, small for gestational age, low birth weight and postpartum hemorrhage).

Another in vitro study will evaluate the immune system contribution in the implantation period and its changes in the different trimesters of pregnancies after ART conception in women with and without adenomyosis. Blood samples will be obtained - Baseline: prior to ovarian stimulation - Post ovarian stimulation (day of HCG, human chorionic gonadotropin, administration) - Post implantation (2 weeks after embryo transfer, the day of first beta HCG measurement -Second (18-24 gestational weeks) and -Third trimester (28-32 gestational week) of eventual subsequent pregnancies).

The aim of this study will be to identify immunological markers such as cellular component and related cytokines in healthy women and women with adenomyosis that undergo ART. In particular the immune system cells population and relative cytokines, the frequency of immune system cells, the interleukins profile, T cells activity and of specific receptors of pregnancy hormone involved in T cell activity will be studied. These results will be linked with estradiol, progesterone and nitric oxide in vivo levels: this will be very important in order to prevent birth losses and to propose new therapies and targets to improve early stages of blastocyst implantation in women with adenomyosis. Forty women with adenomyosis vs. 40 healthy controls will be included in this last part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adenomyosis of the uterus defined with at least one of the following features: (1) heterogeneous myometrium; (2) hypoechoic striation in the myometrium; (3) myometrial anechoic lacunae or cysts; (4) asymmetrical myometrial thickening of the uterine walls.
* Couples who are undergoing a cycle of IVF/ICSI, where a cycle is defined as egg collection following ovarian stimulation.
* First or second IVF or ICSI attempt.
* Absence of severe premature ovarian insufficiency defined by antral follicle count < 8 and AMH (anti-mullerian hormone) < 1ng/ml
* Meet the criteria from the Italian law to be included in a ART program.
* The female partner is ≥18 and < 42 years of age.
* The female partner has a BMI <30.
* Both partners are willing and able to provide written informed consent.

Exclusion Criteria:

* Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within the previous 3 months of study enrolment.
* Other potential causes of implantation failure: in situ leiomyoma, hydrosalpinx, malformed uterus (unicornis, bicornis, septate, duplex), antiphospholipid syndrome
* Uterine fibroids (untreated FIGO, International Federation of Gynecology and Obstetrics, Type 0-I-II and type III-IV fibroids > 3 cm)
* Use of GnRH analogues within previous 3 months.
* Extremely severe male factor infertility (sperm count < 1x 10 6 /ml, use o surgically retrieved spermatozoa)
* Positive plasma viral load for human immunodeficiency virus(HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) for one (or both) in the couple during the year before inclusion
* Couples unable to give fully informed consent to the study.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
live birth after ART | Through study completion, an average of 2 year
  Primary Outcome:Number of live birth after ART attempt defined as delivery of one or more live-born infant at >22 weeks of gestation.

SECONDARY OUTCOMES:
Other ART and pregnancy outcomes | Through study completion, an average of 2 year
  Uterine volume reduction between TV-US measurements at baseline and at time of COH onset
Other ART and pregnancy outcomes | Through study completion, an average of 2 year
  Occurrence of poor responders
Other ART and pregnancy outcomes | Through study completion, an average of 2 year
  Implantation rate
Other ART and pregnancy outcomes | Through study completion, an average of 2 year
  Number of participants with ongoing pregnancy
Other ART and pregnancy outcomes | Immediately after the childbirth
  Preterm delivery rate
Other ART and pregnancy outcomes | Immediately after the childbirth
  Pre-eclampsia occurrence
Other ART and pregnancy outcomes | Immediately after the childbirth
  Caesarean section rate
Other ART and pregnancy outcomes | Immediately after the childbirth
  Fetal malpresentation rate
Other ART and pregnancy outcomes | Immediately after the childbirth
  Small for gestational age rate
Other ART and pregnancy outcomes | Immediately after the childbirth
  Low birth weight (<5 centile) rate
Other ART and pregnancy outcomes | Immediately after the childbirth
  Postpartum hemorrhage(>500 ml) rate

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott JA. Adenomyosis and Abnormal Uterine Bleeding (AUB-A)-Pathogenesis, diagnosis, and management. Best Pract Res Clin Obstet Gynaecol. 2017 Apr;40:68-81. doi: 10.1016/j.bpobgyn.2016.09.006. Epub 2016 Sep 30. PMID 27810281
- [Background] Chapron C, Vannuccini S, Santulli P, Abrao MS, Carmona F, Fraser IS, Gordts S, Guo SW, Just PA, Noel JC, Pistofidis G, Van den Bosch T, Petraglia F. Diagnosing adenomyosis: an integrated clinical and imaging approach. Hum Reprod Update. 2020 Apr 15;26(3):392-411. doi: 10.1093/humupd/dmz049. PMID 32097456
- [Background] Burney RO, Giudice LC. Pathogenesis and pathophysiology of endometriosis. Fertil Steril. 2012 Sep;98(3):511-9. doi: 10.1016/j.fertnstert.2012.06.029. Epub 2012 Jul 20. PMID 22819144
- [Background] Lalani S, Choudhry AJ, Firth B, Bacal V, Walker M, Wen SW, Singh S, Amath A, Hodge M, Chen I. Endometriosis and adverse maternal, fetal and neonatal outcomes, a systematic review and meta-analysis. Hum Reprod. 2018 Oct 1;33(10):1854-1865. doi: 10.1093/humrep/dey269. PMID 30239732
- [Background] Koot YE, van Hooff SR, Boomsma CM, van Leenen D, Groot Koerkamp MJ, Goddijn M, Eijkemans MJ, Fauser BC, Holstege FC, Macklon NS. An endometrial gene expression signature accurately predicts recurrent implantation failure after IVF. Sci Rep. 2016 Jan 22;6:19411. doi: 10.1038/srep19411. PMID 26797113
- [Background] Peng Y et al. Biol Reprod. 2021 Feb 2:ioab017.
- [Background] Nirgianakis K, Kalaitzopoulos DR, Schwartz ASK, Spaanderman M, Kramer BW, Mueller MD, Mueller M. Fertility, pregnancy and neonatal outcomes of patients with adenomyosis: a systematic review and meta-analysis. Reprod Biomed Online. 2021 Jan;42(1):185-206. doi: 10.1016/j.rbmo.2020.09.023. Epub 2020 Oct 4. PMID 33191131
- [Background] Grandi G, Barra F, Ferrero S, Sileo FG, Bertucci E, Napolitano A, Facchinetti F. Hormonal contraception in women with endometriosis: a systematic review. Eur J Contracept Reprod Health Care. 2019 Feb;24(1):61-70. doi: 10.1080/13625187.2018.1550576. Epub 2019 Jan 21. PMID 30664383
- [Background] Grandi G, Mueller MD, Bersinger NA, Facchinetti F, McKinnon BD. The association between progestins, nuclear receptors expression and inflammation in endometrial stromal cells from women with endometriosis. Gynecol Endocrinol. 2017 Sep;33(9):712-715. doi: 10.1080/09513590.2017.1314458. Epub 2017 Apr 17. PMID 28412861
- [Background] Grandi G, Mueller M, Bersinger N, Papadia A, Nirgianakis K, Cagnacci A, McKinnon B. Progestin suppressed inflammation and cell viability of tumor necrosis factor-alpha-stimulated endometriotic stromal cells. Am J Reprod Immunol. 2016 Oct;76(4):292-8. doi: 10.1111/aji.12552. Epub 2016 Aug 12. PMID 27515307
- [Background] Grandi G, Mueller MD, Papadia A, Kocbek V, Bersinger NA, Petraglia F, Cagnacci A, McKinnon B. Inflammation influences steroid hormone receptors targeted by progestins in endometrial stromal cells from women with endometriosis. J Reprod Immunol. 2016 Sep;117:30-8. doi: 10.1016/j.jri.2016.06.004. Epub 2016 Jun 17. PMID 27371899
- [Background] Grandi G, Mueller M, Bersinger NA, Cagnacci A, Volpe A, McKinnon B. Does dienogest influence the inflammatory response of endometriotic cells? A systematic review. Inflamm Res. 2016 Mar;65(3):183-92. doi: 10.1007/s00011-015-0909-7. Epub 2015 Dec 9. PMID 26650031
- [Background] Grandi G, Xholli A, Napolitano A, Palma F, Cagnacci A. Pelvic pain and quality of life of women with endometriosis during quadriphasic estradiol valerate/dienogest oral contraceptive: a patient-preference prospective 24-week pilot study. Reprod Sci. 2015 May;22(5):626-32. doi: 10.1177/1933719114556488. Epub 2014 Nov 13. PMID 25394646
- [Background] Grandi G, Ferrari S, Xholli A, Cannoletta M, Palma F, Romani C, Volpe A, Cagnacci A. Prevalence of menstrual pain in young women: what is dysmenorrhea? J Pain Res. 2012;5:169-74. doi: 10.2147/JPR.S30602. Epub 2012 Jun 20. PMID 22792003
- [Background] Grandi G, Xholli A, Ferrari S, Cannoletta M, Volpe A, Cagnacci A. Intermenstrual pelvic pain, quality of life and mood. Gynecol Obstet Invest. 2013;75(2):97-100. doi: 10.1159/000343997. Epub 2012 Nov 23. PMID 23182853
- [Background] Nirgianakis K, Grandi G, McKinnon B, Bersinger N, Cagnacci A, Mueller M. Dienogest mediates midkine suppression in endometriosis. Hum Reprod. 2016 Sep;31(9):1981-6. doi: 10.1093/humrep/dew180. Epub 2016 Jul 13. PMID 27412246
- [Background] Barra F, Romano A, Grandi G, Facchinetti F, Ferrero S. Future directions in endometriosis treatment: discovery and development of novel inhibitors of estrogen biosynthesis. Expert Opin Investig Drugs. 2019 Jun;28(6):501-504. doi: 10.1080/13543784.2019.1618269. Epub 2019 May 17. No abstract available. PMID 31072144
- [Background] Barra F, Grandi G, Tantari M, Scala C, Facchinetti F, Ferrero S. A comprehensive review of hormonal and biological therapies for endometriosis: latest developments. Expert Opin Biol Ther. 2019 Apr;19(4):343-360. doi: 10.1080/14712598.2019.1581761. Epub 2019 Feb 27. PMID 30763525
- [Background] Kocbek V, Grandi G, Blank F, Wotzkow C, Bersinger NA, Mueller MD, Kyo S, McKinnon BD. TNFalpha-induced IKKbeta complex activation influences epithelial, but not stromal cell survival in endometriosis. Mol Hum Reprod. 2016 Nov;22(11):768-777. doi: 10.1093/molehr/gaw054. Epub 2016 Aug 19. PMID 27542948
- [Background] Cagnacci A, Bellafronte M, Xholli A, Palma F, Carbone MM, Di Carlo C, Grandi G. Impact of laparoscopic cystectomy of endometriotic and non-endometriotic cysts on ovarian volume, antral follicle count (AFC) and ovarian doppler velocimetry. Gynecol Endocrinol. 2016;32(4):298-301. doi: 10.3109/09513590.2016.1142523. Epub 2016 Feb 5. PMID 26850447
- [Background] Pinzauti S, Lazzeri L, Tosti C, Centini G, Orlandini C, Luisi S, Zupi E, Exacoustos C, Petraglia F. Transvaginal sonographic features of diffuse adenomyosis in 18-30-year-old nulligravid women without endometriosis: association with symptoms. Ultrasound Obstet Gynecol. 2015 Dec;46(6):730-6. doi: 10.1002/uog.14834. PMID 25728241
- [Background] Berkhout RP, Lambalk CB, Repping S, Hamer G, Mastenbroek S. Premature expression of the decidualization marker prolactin is associated with repeated implantation failure. Gynecol Endocrinol. 2020 Apr;36(4):360-364. doi: 10.1080/09513590.2019.1650344. Epub 2019 Aug 7. PMID 31389284
- [Background] Berneau SC, Ruane PT, Brison DR, Kimber SJ, Westwood M, Aplin JD. Characterisation of Osteopontin in an In Vitro Model of Embryo Implantation. Cells. 2019 May 9;8(5):432. doi: 10.3390/cells8050432. PMID 31075896
- [Background] Park CW, Choi MH, Yang KM, Song IO. Pregnancy rate in women with adenomyosis undergoing fresh or frozen embryo transfer cycles following gonadotropin-releasing hormone agonist treatment. Clin Exp Reprod Med. 2016 Sep;43(3):169-73. doi: 10.5653/cerm.2016.43.3.169. Epub 2016 Sep 22. PMID 27689040
- [Background] Niu Z, Chen Q, Sun Y, Feng Y. Long-term pituitary downregulation before frozen embryo transfer could improve pregnancy outcomes in women with adenomyosis. Gynecol Endocrinol. 2013 Dec;29(12):1026-30. doi: 10.3109/09513590.2013.824960. Epub 2013 Sep 5. PMID 24006906